CLINICAL TRIAL: NCT05852028
Title: A Real-world Study: Efficacy and Safety of Selinexor-based Regimens for Non-Hodgkin Lymphoma
Brief Title: A Real-world Study of Selinexor-based Regimens for Treatment of Non-Hodgkin Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Other Study IDs: RJ-XLYM-001
Record Dates: First submitted 2023-03-13; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Lymphoma; DLBCL; T Cell Lymphoma
Keywords: SELINEXOR; LYMPHOMA
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell | interventions — selinexor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- selinexor-based regimens: This study is a real-world study to explore the safety and efficacy of selinexor-based therapy in patients with lymphoma. It is planned to enroll 250 patients with lymphoma, including 150 patients with diffuse large B-cell lymphoma and 100 patients with peripheral T and NK/T-cell lymphoma.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — this is a real-world. Patients who use selinexor-based regimens in lymphoma will be followed up without interfering with the choice of treatment options for patients
  Other Names: XPO1 inhibitor

SUMMARY:
This study aims to observe and explore the efficacy and safety of selinexor-based regimen in patients with Non-Hodgkin lymphoma

DETAILED DESCRIPTION:
this study aims to observe and explore the efficacy and safety of selinexor-based regimen in patients with DLBCL or T cell lymphoma. This study is a non-interventional real world, observational study and all registered data are collected from real clinical practice cases. The medical data includes patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, efficacy results and possible prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Know and voluntarily sign the Informed Consent Form (ICF)
* Clinically confirmed DLBCL, T or NK cell lymphoma
* Patients with DLBCL or T or NK cell lymphoma who have used selinexor-based therapy in the past 3 months are included
* Cooperate with clinical diagnosis and treatment management, and provide disease-related past medical history materials

Exclusion Criteria:

* Previously received selinexor
* Poor patient compliance
* physicians evaluate that patients are not suitable for enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DLBCL, T or NK cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | throughout the study, an average of 1 year
  the percentage of patients with complete response and partial response
incidence of adverse events/ serious adverse events | throughout the study, an average of 2 year
  identify patterns of incidence in adverse events

SECONDARY OUTCOMES:
incidence of dose delays or interruptions | throughout the study, an average of 2 year
  calculate incidence and present the occurrence of dose modifying toxicities by cycles and overall

OTHER OUTCOMES:
duration of response (DOR) | throughout the study, an average of 2 year
  DOR is calculated as the time from initial response (complete response or partial response) to date of progression or death, whichever is earlier

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Union Hospital Affiliated to Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided